CLINICAL TRIAL: NCT04894318
Title: The Short Term Beneficıal Effects Of A Low-Fat And Low-Cholesterol Dietary Intervention On LDL Sub-Groups In Dyslipidemic Turkish Patients
Brief Title: The Effect Of Low-Fat And Low-Cholesterol Dietary Intervention On LDL Sub-Groups In Turkısh Dyslipidemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Betül Cicek, Prof.Dr., TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TYL-2018-8497
Record Dates: First submitted 2021-05-05; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia, Low-Fat Low-Cholesterol Diet, LDL Sub-groups
MeSH Terms: conditions — Dyslipidemias | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-fat, low-cholesterol diet (Other): Patients diagnosed with dyslipidemia by the endocrinologist were followed up for 12 weeks with a low-fat, low-cholesterol diet on a monthly basis, provided that they were suitable for each.
  Interventions: Behavioral: Low-fat and low-cholesterol diet

INTERVENTIONS:
Behavioral: Low-fat and low-cholesterol diet — Low-fat (<30% of total energy) and low-cholesterol (<200mg/day) diet total of 12 weeks

SUMMARY:
The aim of this study is to compare LDL sub-group concentration before and after a diet with low-fat and low-cholesterol prescribed to dyslipidemic patients for 12 weeks.

DETAILED DESCRIPTION:
The study was conducted between January 2018-July 2019 in Erciyes University Health Application and Research Center. This study was planned as a clinical trial for treatment and 47 patients were included. All participants were given written consent. The study was evaluated to be ethically appropriate by Erciyes University Faculty of Medicine Clinical Research Ethics Committee.

A low-fat (<30% of total energy), and low-cholesterol (<200 mg/day) diet was planned for the participants at the baseline, according to the gender, lifestyle, working conditions, nutritional habits, BMI, concomitant diseases and risk conditions. The patients were called for monthly controls and followed up for a total of 12 weeks. When the patients admitted at the first and second months, Body Impedance Analyzer (BIA) measurements were performed and dietary adherence was controlled. If necessary, the energy requirements of the patients were re-calculated and their diets were re-newed and if the patients had any questions on the diet, they were answered. Blood samples were taken from the patients at the baseline and after 12 weeks and the effects of a low-fat, low-cholesterol diet on biochemical and anthropometric measurements were evaluated. Energy restricted diet were planed for overweight and obese patients (~ 500-1000 kcal/day). In addition, patients were recommended to walk at a moderate speed for at least 30-40 min per day.

Data Collection A questionnaire including socio-demographic characteristics, nutritional habits, physical activity status, and comorbid diseases was filled by the researcher. The food consumption frequency of the participants was evaluated by dividing the frequencies into four groups as consuming 5-6 times daily, consuming every other day, consuming 1-2 times a week and consuming 1-2 times a month or never at all. Food consumption records were also taken from each patient. Physical activity was questioned by the 'International Physical Activity Questionnaire (short form).

Statistical analysis The suitability of the data for normal distribution was evaluated by histogram, q-q graphs and Shapiro-Wilk test. Variance homogeneity was tested with Levene test. Two groups independent samples t-test and Mann-Whitney U-tests were used for quantitative variables. In the qualitative data, two repeated measurement comparisons were used with McNemar-Bowker test. The paired t-test and Wilcoxon tests were used in the quantitative data for two repeated measurements. Spearman analysis was used to evaluate the relationship between quantitative variables. Data analysis was performed by Turcosa Cloud (Turcosa Ltd Co) statistical software. Significance level was accepted as p<0.05.

Anthropometric measurements After the completing the questionnaire, anthropometric measurements were taken. Body weight: When the patient was in fasting state in the morning measured with thin clothes. While measuring body weight, the individual was asked to remove his heavy clothes (coats, jackets, etc.), belongings in the pockets (wallet, key ring, phone, address book etc.) and shoes. Attention is given to place the feet on the balance and to ensure a balanced distribution of body weight to the two feet. The individual was asked to stand upright and without moving. The measurement was made with a sensitivity of 0.1 kg (100 g). Height: The height was measured with a stadiometer while the feet were side-by-side and the head was in the Frankfort plane. Body mass index (BMI): BMI was calculated by dividing subjects body weight by square of his/her height. [BMI = Body weight (kg)/height (m)²]. Waist circumference: The waist circumference was measured with a non-elastic tape measuring the mid-point between the lower rib and the crista iliac crest. Waist-to height ratio: It was calculated by the division of waist circumference (cm) into height (cm). Neck circumference: Neck circumference was measured with a non-elastic plastic band from the middle of the neck height between the middle cervical spine and the middle anterior neck with a sensitivity of 0.1 cm. In men with Adam's apple, it was measured just below the protrusion. BIA measurements: Body composition of the participants was determined with Tanita BC-418 MA (Tanita Corporation of America, Inc., Arlington Heights, IL) device. In order to make accurate measurements; metal jewelery on individuals, socks, clothes that will affect the measurement excessively were removed and information about the person's age, height, gender and whether they are dealing with regular sports activities were entered into the device. Then, individuals were removed from the instrument with their heels on the electrodes and the measurement was made. It was taken into consideration that participants did not perform intensive physical activity 24-48 hours before the measurement. It was observed that individuals did not have heavy physical activity 24-48 hours before the measurement, they were fasted for at least 4 hours, no alcohol was used 24 hours before, and they did not consume too much beverages (tea, coffee) before the measurement (at least 4 hours).

Biochemical parameters In the Endocrinology polyclinic; the patients were diagnosed with dyslipidemia by an endocrinologist and their fasting blood glucose (mg/dL), triglycerides (mg/dL), total cholesterol (mg/dL), HDL-cholesterol (mg/dL), LDL-cholesterol (mg/dL) levels were evaluated. Patients were selected according to the inclusion criteria and blood was drawn after fasting for at least 10-12 hours. Very low density lipoprotein (VLDL (mg/dL)), large-LDL (mg/dL), small-LDL (mg/dL) medium density lipoprotein (IDL (mg/dL)) (Mid A, B, C) values. After centrifugation, blood samples were kept in the freezer at -80°C in Erciyes University Endocrinology Service until analysis period. For patients who were not initially evaluated for insulin (mg/dL), some blood was collected and delivered to Erciyes University Blood Collection Department and studied at the Central Biochemistry Laboratory of Erciyes University. Fasting blood glucose, triglyceride, total cholesterol, HDL-cholesterol and LDL-cholesterol levels were measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland). Insulin was measured by the ECLIA study method using the Roche Diagnostics (Mannheim, Germany). LDL subgroups were measured in serum samples using a Lipoprint System (Quantimetrix Inc., Redondo Beach, CA, USA). This system separates lipoproteins in a non-denaturing gel gradient of polyacrylamide based on net surface charge and size. The dye binds proportionally to the relative amount of cholesterol in each lipoprotein. After the electrophoresis, densitometric analyzes and proportional concentrations of lipoprotein classes and subclasses were calculated on the Lipoware software. In this system, VLDL, IDL corresponding to 3 midbands (Mid A, B, C) and 7 LDL subgroups: LDL-1 to -2 (large, bouyant, pattern A); LDL-3 to -7 (small, dense; pattern B). The system also gives the average LDL particle size. Type A if particle size was ≥268Â, medium level if particle size was 265-268Â, type B if particle size was ≤265Â.

ELIGIBILITY:
Inclusion Criteria

* Being diagnosed with dyslipidemia by an endocrinologist
* Those who do not have a history of diabetes, hyperthyroidism, hypothyroidism (including those who have hypothyroidism but receive replacement therapy)
* 25-65 years
* Body Mass Index (BMI) = 25-40 kg/m²
* Smoking three or less than three cigarettes a day
* Not using herbal supplements.
* Not being in pregnancy or lactation period
* Volunteering to participate in the study

Exclusion Criteria:

* Not being diagnosed with dyslipidemia
* Using a drug that affects the lipid profile
* Not being in the age range of 25-65
* BMI = 25-40 kg/m² not
* Smoking more than three cigarettes a day
* Using herbal supplements
* Being in the pregnancy or lactation period
* Not willing to participate in the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Baseline LDL subgroups at 12 weeks | Baseline and 12 weeks
  LDL subgroups were measured in serum samples using a Lipoprint System (Quantimetrix Inc., Redondo Beach, CA, USA). This system separates lipoproteins in a non-denaturing gel gradient of polyacrylamide based on net surface charge and size. The dye binds proportionally to the relative amount of cholesterol in each lipoprotein. After the electrophoresis, densitometric analyzes and proportional concentrations of lipoprotein classes and subclasses were calculated on the Lipoware software. In this system, VLDL, IDL corresponding to 3 midbands (Mid A, B, C) and 7 LDL subgroups: LDL-1 to -2 (large, bouyant, pattern A); LDL-3 to -7 (small, dense; pattern B). The system also gives the average LDL particle size. Type A if particle size was ≥268Â, medium level if particle size was 265-268Â, type B if particle size was ≤265Â

SECONDARY OUTCOMES:
Change in Baseline body weight at 12 weeks | Baseline and 12 weeks
  Body weight in kilograms
Change in Baseline height at 12 weeks | Baseline and 12 weeks
  Height in centimeter
Change in Baseline Body mass index (BMI) at 12 weeks | Baseline and 12 weeks
  Body mass index (BMI) was calculated by dividing subjects body weight by square of his/her height. [BMI = Body weight (kg)/height (m)²]
Change in Baseline waist circumference at 12 weeks | Baseline and 12 weeks
  Waist circumference in centimeter
Change in Baseline waist-to-height ratio at 12 weeks | Baseline and 12 weeks
  Waist-to-height ratio was calculated by the division of waist circumference (cm) into height (cm)
Change in Baseline neck circumference at 12 weeks | Baseline and 12 weeks
  Neck circumference in centimeter
Change in Baseline fat percentage at 12 weeks | Baseline and 12 weeks
  Fat percentage (%) was measured by Tanita BC-418 MA (Tanita Corporation of America, Inc., Arlington Heights, IL)
Change in Baseline muscle mass at 12 weeks | Baseline and 12 weeks
  Muscle mass was measured by Tanita BC-418 MA (Tanita Corporation of America, Inc., Arlington Heights, IL)
Change in Baseline blood sugar at 12 weeks | Baseline and 12 weeks
  Blood sugar (mg/dL) was measured after at least 10-12 hours of fasting. Fasting blood glucose was measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland).
Change in Baseline triglycerides at 12 weeks | Baseline and 12 weeks
  Triglycerides (mg/dL) was measured after at least 10-12 hours of fasting. Triglyceride was measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland). Triglycerides measurement is used in the diagnosis of dyslipidemia and the risk of cardiovascular disease increases above 150 mg/dL.
Change in Baseline total cholesterol at 12 weeks | Baseline and 12 weeks
  Total cholesterol (mg/dL) was measured after at least 10-12 hours of fasting. Total cholesterol was measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland). Total cholesterol measurement is used in the diagnosis of dyslipidemia and the risk of cardiovascular disease increases above 200 mg/dL.
Change in Baseline HDL-cholesterol at 12 weeks | Baseline and 12 weeks
  HDL-cholesterol (mg/dL) was measured after at least 10-12 hours of fasting. HDL-cholesterol was measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland). HDL cholesterol measurement is used in the diagnosis of dyslipidemia and the increase in HDL cholesterol reduces the risk of cardiovascular disease.
Change in Baseline LDL-cholesterol at 12 weeks | Baseline and 12 weeks
  LDL-cholesterol (mg/dL) was measured after at least 10-12 hours of fasting. LDL-cholesterol levels was measured by spectrophotometric method using Roche Diagnostics (Basel, Switzerland). LDL-cholesterol measurement is used in the diagnosis of dyslipidemia and the risk of cardiovascular disease increases above 130 mg/dL.
Change in Baseline insulin at 12 weeks | Baseline and 12 weeks
  LDL-cholesterol (mg/dL) was measured after at least 10-12 hours of fasting. Insulin was measured by the ECLIA study method using the Roche Diagnostics (Mannheim, Germany).
Change in Baseline blood pressure Levels at 12 weeks | Baseline and 12 weeks
  Blood pressure was measured with a device called a sphygmomanometer while patients were at rest. High blood pressure is one of the most important risk factors for cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ülger Kaçar Mutlutürk, Phd, Principal Investigator — TC Erciyes University; Fahri Bayram, Prof.Dr., Study Director — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All off the individual
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the date

REFERENCES:
- [Result] Jellinger PS, Smith DA, Mehta AE, Ganda O, Handelsman Y, Rodbard HW, Shepherd MD, Seibel JA; AACE Task Force for Management of Dyslipidemia and Prevention of Atherosclerosis. American Association of Clinical Endocrinologists' Guidelines for Management of Dyslipidemia and Prevention of Atherosclerosis. Endocr Pract. 2012 Mar-Apr;18 Suppl 1:1-78. doi: 10.4158/ep.18.s1.1. No abstract available. PMID 22522068
- [Result] Bayram F, Kocer D, Gundogan K, Kaya A, Demir O, Coskun R, Sabuncu T, Karaman A, Cesur M, Rizzo M, Toth PP, Gedik V. Prevalence of dyslipidemia and associated risk factors in Turkish adults. J Clin Lipidol. 2014 Mar-Apr;8(2):206-16. doi: 10.1016/j.jacl.2013.12.011. Epub 2014 Jan 19. PMID 24636181
- [Result] Mahley RW, Pepin J, Palaoglu KE, Malloy MJ, Kane JP, Bersot TP. Low levels of high density lipoproteins in Turks, a population with elevated hepatic lipase. High density lipoprotein characterization and gender-specific effects of apolipoprotein e genotype. J Lipid Res. 2000 Aug;41(8):1290-301. PMID 10946017
- [Result] Bedard A, Corneau L, Lamarche B, Dodin S, Lemieux S. Sex Differences in the Impact of the Mediterranean Diet on LDL Particle Size Distribution and Oxidation. Nutrients. 2015 May 15;7(5):3705-23. doi: 10.3390/nu7053705. PMID 25988764
- [Result] El Harchaoui K, van der Steeg WA, Stroes ES, Kuivenhoven JA, Otvos JD, Wareham NJ, Hutten BA, Kastelein JJ, Khaw KT, Boekholdt SM. Value of low-density lipoprotein particle number and size as predictors of coronary artery disease in apparently healthy men and women: the EPIC-Norfolk Prospective Population Study. J Am Coll Cardiol. 2007 Feb 6;49(5):547-53. doi: 10.1016/j.jacc.2006.09.043. Epub 2007 Jan 22. PMID 17276177
- [Result] Ai M, Otokozawa S, Asztalos BF, Ito Y, Nakajima K, White CC, Cupples LA, Wilson PW, Schaefer EJ. Small dense LDL cholesterol and coronary heart disease: results from the Framingham Offspring Study. Clin Chem. 2010 Jun;56(6):967-76. doi: 10.1373/clinchem.2009.137489. Epub 2010 Apr 29. PMID 20431054
- [Result] Gerber PA, Nikolic D, Rizzo M. Small, dense LDL: an update. Curr Opin Cardiol. 2017 Jul;32(4):454-459. doi: 10.1097/HCO.0000000000000410. PMID 28426445
- [Result] Feingold KR. Introduction to Lipids and Lipoproteins. 2024 Jan 14. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK305896/ PMID 26247089
- [Result] Ivanova EA, Myasoedova VA, Melnichenko AA, Grechko AV, Orekhov AN. Small Dense Low-Density Lipoprotein as Biomarker for Atherosclerotic Diseases. Oxid Med Cell Longev. 2017;2017:1273042. doi: 10.1155/2017/1273042. Epub 2017 May 7. PMID 28572872
- [Result] Guay V, Lamarche B, Charest A, Tremblay AJ, Couture P. Effect of short-term low- and high-fat diets on low-density lipoprotein particle size in normolipidemic subjects. Metabolism. 2012 Jan;61(1):76-83. doi: 10.1016/j.metabol.2011.06.002. Epub 2011 Aug 3. PMID 21816443
- [Result] Authors/Task Force Members; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2019 ESC/EAS guidelines for the management of dyslipidaemias: Lipid modification to reduce cardiovascular risk. Atherosclerosis. 2019 Nov;290:140-205. doi: 10.1016/j.atherosclerosis.2019.08.014. Epub 2019 Aug 31. No abstract available. PMID 31591002
- [Result] Schwingshackl L, Hoffmann G. Comparison of effects of long-term low-fat vs high-fat diets on blood lipid levels in overweight or obese patients: a systematic review and meta-analysis. J Acad Nutr Diet. 2013 Dec;113(12):1640-61. doi: 10.1016/j.jand.2013.07.010. Epub 2013 Oct 17. PMID 24139973
- [Result] Wu L, Ma D, Walton-Moss B, He Z. Effects of low-fat diet on serum lipids in premenopausal and postmenopausal women: a meta-analysis of randomized controlled trials. Menopause. 2014 Jan;21(1):89-99. doi: 10.1097/GME.0b013e318291f5c2. PMID 23736858
- [Result] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Result] Zen V, Fuchs FD, Wainstein MV, Goncalves SC, Biavatti K, Riedner CE, Fuchs FC, Wainstein RV, Rhoden EL, Ribeiro JP, Fuchs SC. Neck circumference and central obesity are independent predictors of coronary artery disease in patients undergoing coronary angiography. Am J Cardiovasc Dis. 2012;2(4):323-30. Epub 2012 Oct 25. PMID 23173107
- [Result] Hoefner DM, Hodel SD, O'Brien JF, Branum EL, Sun D, Meissner I, McConnell JP. Development of a rapid, quantitative method for LDL subfractionation with use of the Quantimetrix Lipoprint LDL System. Clin Chem. 2001 Feb;47(2):266-74. PMID 11159775
- [Result] Kostis JB. The importance of managing hypertension and dyslipidemia to decrease cardiovascular disease. Cardiovasc Drugs Ther. 2007 Aug;21(4):297-309. doi: 10.1007/s10557-007-6032-4. PMID 17605096
- [Result] Aoki T, Yagi H, Sumino H, Tsunekawa K, Araki O, Kimura T, Nara M, Ogiwara T, Nakajima K, Murakami M. Relationship between carotid artery intima-media thickness and small dense low-density lipoprotein cholesterol concentrations measured by homogenous assay in Japanese subjects. Clin Chim Acta. 2015 Mar 10;442:110-4. doi: 10.1016/j.cca.2015.01.010. Epub 2015 Jan 17. PMID 25603407
- [Result] Taylan E, Tuncel EP. Distribution of LDL subgroups in patients with hyperlipidemia. Turk J Med Sci. 2016 Feb 17;46(2):374-80. doi: 10.3906/sag-1410-40. PMID 27511499
- [Result] Jacobson TA, Maki KC, Orringer CE, Jones PH, Kris-Etherton P, Sikand G, La Forge R, Daniels SR, Wilson DP, Morris PB, Wild RA, Grundy SM, Daviglus M, Ferdinand KC, Vijayaraghavan K, Deedwania PC, Aberg JA, Liao KP, McKenney JM, Ross JL, Braun LT, Ito MK, Bays HE, Brown WV, Underberg JA; NLA Expert Panel. National Lipid Association Recommendations for Patient-Centered Management of Dyslipidemia: Part 2. J Clin Lipidol. 2015 Nov-Dec;9(6 Suppl):S1-122.e1. doi: 10.1016/j.jacl.2015.09.002. Epub 2015 Sep 18. PMID 26699442
- [Result] Zhu Z, Wu F, Lu Y, Wang Z, Zang J, Yu H, Guo C, Jia X, Shen X, Ding G. The Association of Dietary Cholesterol and Fatty Acids with Dyslipidemia in Chinese Metropolitan Men and Women. Nutrients. 2018 Jul 25;10(8):961. doi: 10.3390/nu10080961. PMID 30044444
- [Result] Ensign W, Hill N, Heward CB. Disparate LDL phenotypic classification among 4 different methods assessing LDL particle characteristics. Clin Chem. 2006 Sep;52(9):1722-7. doi: 10.1373/clinchem.2005.059949. Epub 2006 Jun 1. PMID 16740651
- [Result] Ohmura H, Mokuno H, Sawano M, Hatsumi C, Mitsugi Y, Watanabe Y, Daida H, Yamaguchi H. Lipid compositional differences of small, dense low-density lipoprotein particle influence its oxidative susceptibility: possible implication of increased risk of coronary artery disease in subjects with phenotype B. Metabolism. 2002 Sep;51(9):1081-7. doi: 10.1053/meta.2002.34695. PMID 12200749
- [Result] Chiu S, Williams PT, Krauss RM. Effects of a very high saturated fat diet on LDL particles in adults with atherogenic dyslipidemia: A randomized controlled trial. PLoS One. 2017 Feb 6;12(2):e0170664. doi: 10.1371/journal.pone.0170664. eCollection 2017. PMID 28166253
- [Result] Hosaka S, Okada Y, Maruyama K, Maruyama D. Increased intima-media thickness of the carotid artery in Japanese female type 2 diabetic patients with 'midband lipoprotein'. Diabetes Res Clin Pract. 2007 Mar;75(3):333-8. doi: 10.1016/j.diabres.2006.07.032. Epub 2006 Sep 8. PMID 16963151
- [Result] Srisawasdi P, Vanavanan S, Rochanawutanon M, Pornsuriyasak P, Tantrakul V, Kruthkul K, Kotani K. Heterogeneous properties of intermediate- and low-density lipoprotein subpopulations. Clin Biochem. 2013 Oct;46(15):1509-15. doi: 10.1016/j.clinbiochem.2013.06.021. Epub 2013 Jul 2. PMID 23830843
- [Result] Klop B, Elte JW, Cabezas MC. Dyslipidemia in obesity: mechanisms and potential targets. Nutrients. 2013 Apr 12;5(4):1218-40. doi: 10.3390/nu5041218. PMID 23584084
- [Result] Taylor AE, Ebrahim S, Ben-Shlomo Y, Martin RM, Whincup PH, Yarnell JW, Wannamethee SG, Lawlor DA. Comparison of the associations of body mass index and measures of central adiposity and fat mass with coronary heart disease, diabetes, and all-cause mortality: a study using data from 4 UK cohorts. Am J Clin Nutr. 2010 Mar;91(3):547-56. doi: 10.3945/ajcn.2009.28757. Epub 2010 Jan 20. PMID 20089729
- [Result] Frimel TN, Sinacore DR, Villareal DT. Exercise attenuates the weight-loss-induced reduction in muscle mass in frail obese older adults. Med Sci Sports Exerc. 2008 Jul;40(7):1213-9. doi: 10.1249/MSS.0b013e31816a85ce. PMID 18580399
- [Result] Newman AB, Lee JS, Visser M, Goodpaster BH, Kritchevsky SB, Tylavsky FA, Nevitt M, Harris TB. Weight change and the conservation of lean mass in old age: the Health, Aging and Body Composition Study. Am J Clin Nutr. 2005 Oct;82(4):872-8; quiz 915-6. doi: 10.1093/ajcn/82.4.872. PMID 16210719
- [Result] Yang XP, Reckelhoff JF. Estrogen, hormonal replacement therapy and cardiovascular disease. Curr Opin Nephrol Hypertens. 2011 Mar;20(2):133-8. doi: 10.1097/MNH.0b013e3283431921. PMID 21178615
- [Result] Pai JK, Manson JE. Acceleration of cardiovascular risk during the late menopausal transition. Menopause. 2013 Jan;20(1):1-2. doi: 10.1097/gme.0b013e318278e9b4. No abstract available. PMID 23266836
- [Result] Stock EO, Redberg R. Cardiovascular disease in women. Curr Probl Cardiol. 2012 Nov;37(11):450-526. doi: 10.1016/j.cpcardiol.2012.07.001. PMID 23047015
- See also: TEMD Obezite, Dislipidemi, Hipertansiyon Çalışma Grubu' TEMD Dislipidemi Tanı ve Tedavi Kılavuzu', Ankara, Nisan 2019: 13-40 (in Turkish) — http://www.temd.org.tr/admin/uploads/tbl_gruplar/20200930134854-2020tbl_gruplar513182565d.pdf
- See also: Türkiye Beslenme Rehberi TUBER 2015, T.C. Saglık Bakanlıgı Yayın No: 1031, Ankara 2016.Erisim:[https://dosyasb.saglik.gov.tr/Eklenti/10915,tuberturkiyebeslenme-rehberipdf.pdf], Date of access: 18.10.2018 (in Turkish). — https://dosyasb.saglik.gov.tr/Eklenti/10915,tuber-turkiye-beslenme-rehberipdf.pdf